CLINICAL TRIAL: NCT04263662
Title: Implementation of a New Analgesia-sedation Algorithm in the Pediatric Intensive Care Unit to Reduce Overall Benzodiazepine Usage
Brief Title: Implementation of an Analgesia-sedation Algorithm in the Pediatric ICU to Reduce Benzodiazepine Use
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Nilesh M. Mehta, Professor of Anaesthesia, Critical Care, Harvard Medical School, Boston Children's Hospital
Other Study IDs: IRB-P00032707
Record Dates: First submitted 2020-02-05; First posted 2020-02-11 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Mechanical Ventilation; Sedation
Keywords: Analgesia; Sedation; Dexmedetomidine; Mechanical Ventilation; Delirium
MeSH Terms: conditions — Agnosia; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-algorithm: Patients admitted to the pediatric ICU who are intubated for greater than 24 hours prior to implementation of an analgesia-sedation algorithm.
- Post-algorithm: Patients admitted to the pediatric ICU who are intubated for greater than 24 hours after implementation of an analgesia-sedation algorithm.
  Interventions: Other: Analgesia-Sedation algorithm

INTERVENTIONS:
Other: Analgesia-Sedation algorithm — The analgesia-sedation algorithm is a suggested protocol for approach to providing analgesia and sedation to patients admitted to the pediatric ICU who are newly intubated. The approach focuses on using dexmedetomidine as the primary sedative, non-opioids as the primary analgesia, then stepwise approach to adding in adjunctives (e.g. opioids, non-benzodiazepines) with the intention of minimizing benzodiazepine exposure and utilizing minimal-dose effective analgesia/sedative dosing.
  Groups: Post-algorithm

SUMMARY:
The purpose of the study is to develop and implement an evidence-based analgesia-sedation algorithm in the pediatric intensive care unit (PICU) using quality improvement and implementation science methodology. The analgesia-sedation protocol will be implemented for patients admitted to the pediatric ICU who require mechanical ventilation for greater than 24 hours. Specifically, we will examine the impact of this implementation on total benzodiazepine usage, ICU length of stay, and ventilator free days, using a pre- and post- algorithm implementation comparative design.

DETAILED DESCRIPTION:
Study Design and exposures:

1. Development of an evidence-based analgesia-sedation algorithm for mechanically ventilated children using an iterative, multidisciplinary collaborative effort.
2. Exposure: Implementation of the analgesia-sedation algorithm using standard quality improvement (QI) methodology. This will include education, awareness, wash-in phases followed by actual implementation with support. We will use a before-after comparison design.

Patients will be eligible if they are admitted to the medical and multidisciplinary (medical/surgical) ICUs at Boston Children's Hospital and require mechanical ventilatory support for greater than 24 hours.

Study period: Eligible patients who are admitted to the ICUs between August 1st 2017 - February 28th 2018 (pre-implementation) and August 1st 2019 - February 28th 2020 (post-implementation) will be enrolled.

Data collection: Retrospective chart review, with manual data entry in REDCap. Pre-intervention data will be collected starting July 2019. After the intervention begins in July 2019, data collection will occur monthly with the intent of collecting compliance data through analyzing usage of a new electronic medical record order set designed specifically for this intervention and feeding that back to staff members via electronic communication and meeting presentations in order to assess barriers to implementation of the new algorithm. Prospective post-intervention data collection will begin in September 2019 and end in March 2020.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the pediatric ICU between August 1st 2017 - February 28th 2018 and August 1st 2019 - February 28th 2020
* Intubated for greater than 24 hours will be eligible

Exclusion Criteria:

* Ventilated via a tracheostomy at the time of admission
* Pre-admission documentation of dexmedetomidine allergy
* Receiving a midazolam infusion for greater than 4 hours at the time of admission
* Admitted to the ICU for initiation of the rapid-escalation midazolam protocol for status epilepticus

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients admitted to the ICU who receive invasive mechanical ventilation via an endotracheal or nasotracheal tube and are potentially eligible to follow the analgesia-sedation algorithm.
Sampling Method: Non-Probability Sample
Enrollment: 680 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Benzodiazepine exposure | We will collect data (after hospital discharge) on amount of benzodiazepine administration in their ICU stay for each ICU patient admitted between Aug 2017 - Feb 2018 (pre-intervention group), and Aug 2019 - Feb 2020 (post-intervention group).
  Total exposure of benzodiazepines (midazolam, lorazepam, diazepam) measured per kilogram of weight over the patient's duration of ICU stay.

SECONDARY OUTCOMES:
Opioid exposure | We will collect data (after hospital discharge) on amount of opioid administration in their ICU stay for each ICU patient admitted between Aug 2017 - Feb 2018 (pre-intervention group), and Aug 2019 - Feb 2020 (post-intervention group).
  Total exposure of opioids (measured in morphine equivalents) measured per kilogram of weight over the patient's duration of ICU stay.
ICU length of stay | We will collect data (after hospital discharge) on duration of ICU stay for each ICU patient admitted between Aug 2017 - Feb 2018 (pre-intervention group), and Aug 2019 - Feb 2020 (post-intervention group).
  Duration of stay in the ICU measured in days
Ventilator free days | We will collect data (after hospital discharge) on duration of intubation for each ICU patient admitted between Aug 2017 - Feb 2018 (pre-intervention group), and Aug 2019 - Feb 2020 (post-intervention group).
  Duration of time off of invasive mechanical ventilation during the ICU stay
Adverse events | We will collect data (after hospital discharge) on morbidity events for each ICU patient admitted between Aug 2017 - Feb 2018 (pre-intervention group), and Aug 2019 - Feb 2020 (post-intervention group).
  Frequency of morbidities, e.g. unplanned extubation, failed extubation, cardiorespiratory arrest events, unintentional dislodgment of other lines/tubes, re-admission to the hospital/ICU within 24 hours of discharge/transfer.
State behavioral scale (SBS) scores | We will collect data (after hospital discharge) on documented SBS scores for each ICU patient admitted between Aug 2017 - Feb 2018 (pre-intervention group), and Aug 2019 - Feb 2020 (post-intervention group).
  Difference between the desired SBS score and the recorded SBS score
Cornell Assessment of Pediatric Delirium (CAPD) scores | We will collect data (after hospital discharge) on documented CAPD scores for each ICU patient admitted between Aug 2019 - Feb 2020 (post-intervention group only).
  CAPD scores for patients during their ICU stay

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No